CLINICAL TRIAL: NCT05253066
Title: An Open, Multicenter, Randomized Controlled Clinical Study of Chidamide Combined With Exemestane (+/- Goserelin) Versus Neoadjuvant Chemotherapy in Patients of Stage II-III HR-positive/HER2-negative Breast Cancer
Brief Title: Chidamide Combined With Exemestane (+/- Goserelin) Versus Neoadjuvant Chemotherapy in Patients of Stage II-III HR-positive/HER2-negative Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Director, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUKDEN5
Record Dates: First submitted 2022-01-13; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Goserelin; Drug Therapy; Docetaxel; Epirubicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chidamide group (Experimental): Chidamide combined with exemestane (+/- goserelin)
  Interventions: Drug: Chidamide combined with exemestane (+/- goserelin)
- chemotherapy group (Active Comparator): Chemotherapy with docetaxel plus epirubicin or change of chemotherapy regimen (at the discretion of the clinician)
  Interventions: Drug: Chemotherapy with docetaxel plus epirubicin or change of chemotherapy regimen (at the discretion of the clinician)

INTERVENTIONS:
Drug: Chidamide combined with exemestane (+/- goserelin) — Chidamide combined with exemestane (+/- goserelin)
  Arms: Chidamide group
Drug: Chemotherapy with docetaxel plus epirubicin or change of chemotherapy regimen (at the discretion of the clinician) — Chemotherapy with docetaxel plus epirubicin or change of chemotherapy regimen (at the discretion of the clinician)
  Arms: chemotherapy group

SUMMARY:
This is an open, multicenter, randomized controlled clinical study aimed to explore the efficacy and safety of chidamide combined with exemestane (+/- goserelin) versus chemotherapy in the neoadjuvant treatment of stage II-III HR +/HER2- breast cancer patients with poor response to previous chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* female patients aged greater than or equal to 18 years and less than or equal to 75 years, meet one of the following:

  1. previous oophorectomy, or age ≥ 60 years;
  2. age < 60 years, natural postmenopausal status (defined as at least 12 consecutive months of spontaneous cessation of regular menstruation, and no other pathological or physiological causes), E2 and FSH in postmenopausal levels;
  3. premenopausal or perimenopausal female patients, must be willing to receive LHRH agonist therapy during the study;
* all patients were confirmed by histopathology as estrogen receptor (ER) positive (> 10%), HER2 receptor negative.Follow the 2018 version of ASCO-CAP HER2-negative interpretation guideline criteria;
* tumor stage II-III meeting the AJCC 8th version criteria, patients who have previously received 2 cycles of TE regimen chemotherapy, with disease evaluation of SD or PD;
* KPS score ≥ 70 points;
* organ function level must meet the following requirements:

  1. bone marrow function ANC ≥ 1.5 × 109/L (14 without growth factors); PLT ≥ 100 × 109/L (7 without corrective treatment); Hb ≥ 100 g/L (7) without corrective treatment;
  2. liver and kidney function TBIL ≤ 1.5 × ULN; ALT and AST ≤ 3 × ULN; BUN and Cr ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula);
* able to undergo needle biopsy;
* voluntarily join this study, sign informed consent, have good compliance and are willing to cooperate with follow-up

Exclusion Criteria:

* received any form of anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.);
* received any other anti-tumor therapy at the same time;
* breast cancer, inflammatory breast cancer or occult breast cancer;
* stage IV breast cancer;
* breast cancer without histopathological diagnosis;

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-02-25 (Estimated); Primary Completion 2022-07-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to approximately 48 months

SECONDARY OUTCOMES:
pCR：Upon completion of neoadjuvant therapy and surgery, there was no residual invasive carcinoma present in the pathologic assessment of the resected breast cancer samples stained with hematoxylin and eosin and all ipsilateral lymph node samples. | Up to approximately 48 months
Residual tumor burden (RCB) classification | Up to approximately 48 months
Total breast pathological complete remission rate (bpCR) | Up to approximately 48 months
PEPI classification | Up to approximately 48 months
Breast-conserving rate | Up to approximately 48 months
patient-reported outcome（PRO）：evaluate daily functioning and health outcomes from the patient's perspective by HRQOL | Up to approximately 48 months
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Up to approximately 48 months
Number of participants with treatment-related serious adverse event as assessed by CTCAE v5.0 | Up to approximately 48 months